CLINICAL TRIAL: NCT01509872
Title: An RCT Comparing Trauma-Focused Cognitive Behavioral Therapy (a Specific Psychological Intervention) and A Child Friendly Space (a Non-trauma Focused Psychosocial Intervention) in Reducing Psychological Distress Among War-affected Children
Brief Title: Psychological and Psychosocial Intervention With War-Affected Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Transcultural Psychosocial Organization Nepal (Other); UNICEF (Other)
Responsible Party: Principal Investigator, Paul O'Callaghan, Principal Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PREC73-2011
Record Dates: First submitted 2012-01-06; First posted 2012-01-13 (Estimated); Results first posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Stress Disorders, Post-Traumatic; Depression; Anxiety; Conduct; Pro-social Behavior
Keywords: Trauma-Focused Cognitive Behavior Therapy; War-affected Children; Post-traumatic Stress Symptoms; Psychosocial Distress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Behavior

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trauma-Focused Cognitive Behavioral Therapy (Experimental): Trauma-Focused Cognitive Behaviour Therapy (Cohen, Mannarino, Deblinger, 2006; Smith and Saunders, 2005) is a child-friendly, manualised psychological intervention for children who experience nightmares, flashbacks, anxiety, anger, social isolation, poor concentration or self-blame after experiencing or witnessing a violent and terrifying life event (e.g. rape, murder, abduction etc). This intervention was culturally modified for use with war-affected children.
  Interventions: Behavioral: Trauma Focused Cognitive Behavioral Therapy
- A Child Friendly Space (Active Comparator): A Child Friendly Space is a psychosocial intervention combining creative (e.g. art), imaginative (e.g. drama), physical (e.g. football), communicative (e.g. group discussions) and manipulative activities (e.g. story telling). It aids children's natural development by providing a safe place for children to learn, express themselves, grow and develop, supported by trained animators and peer educators.
  Interventions: Behavioral: Child Friendly Space

INTERVENTIONS:
Behavioral: Trauma Focused Cognitive Behavioral Therapy — 9 sessions of manualised, culturally modified, group-based trauma-focused cognitive behavioral therapy
  Arms: Trauma-Focused Cognitive Behavioral Therapy
Behavioral: Child Friendly Space — 9 sessions of a manualised, culturally appropriate, non trauma-focused psychosocial intervention
  Arms: A Child Friendly Space

SUMMARY:
The investigators are interested in knowing whether a group-based, trauma-focused intervention (Trauma Focused Cognitive Behavioral Therapy) is superior to a more general, non trauma-focused, psychosocial intervention (Child Friendly Spaces) in reducing post-traumatic stress, depression and anxiety and conduct problems and increasing pro-social behavior among war-affected children in the Democratic Republic of Congo.

ELIGIBILITY:
Inclusion Criteria:

* under 18 years of age,
* witness to a violent event involving a real or perceived direct threat to life,
* ability to attend a 3-week intervention

Exclusion Criteria:

* psychosis,
* mental retardation,
* inability to understand Swahili,
* severe emotional & behavioral problems that made group participation impossible

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ciarán Shannon, BA, MA, DClin, Study Director — British Psychological Society (Chartered Clinical Psychologist)
Locations (1):
- Child Friendly Space, Mwenga, South Kivu, Republic of the Congo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trauma-Focused Cognitive Behavioral Therapy | A Child Friendly Space
Started | 26 | 24
Post-Intervention Assessment | 26 | 24
Completed | 25 | 24
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trauma-Focused Cognitive Behavioral Therapy | A Child Friendly Space | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.77 (1.58) | 15.00 (1.64) | 14.88 (1.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 16 | 11 | 27
Region of Enrollment [Number; unit: participants]
  Congo, The Democratic Republic of the | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-traumatic Stress Symptoms as Measured by the University of California Los Angelus Post Traumatic Stress Disorder -Reaction Index
Description: The UCLA PTSD Reaction Index is a self-report questionnaire that measures exposure to traumatic events and assesses post-tramatic stress symptoms in school-age children and adolescents. The Congolese Swahili version used in the study had 22 items and assesses the frequency of occurrence of PTSD symptoms during the past week (rated from 0 = none of the time to 4 = most of the time). The scale ranged from 0 (no symptoms) to 88 (highest score possible). Although no cut-off score was used, the higher the score of the scale the higher the number of PTSD symptoms experienced.
Time Frame: baseline, 3 week post-intervention and 6-month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trauma-Focused Cognitive Behavioral Therapy | A Child Friendly Space
Number analyzed (Participants) | 26 | 24
units on a scale
  Pre-Intervention Scores | 47.77 (6.62) | 45.79 (6.87)
  Post-Intervention Scores | 21.54 (10.13) | 21.13 (6.95)
  6 month Follow-Up Intervention Scores | 18.42 (6.17) | 15.88 (7.03)

2. Secondary Outcome: Change in Internalizing Symptoms as Measured by the African Youth Psychosocial Assessment Instrument
Description: The African Youth Psychosocial Assessment Instrument is a self-report questionnaire that measures internalizing, externalizing, conduct and pro-social (daily life functioning) skills symptoms. The Congolese Swahili version of the AYPA contained 19 questions on internalizing symptoms and assesses the frequency of occurrence of internalizing symptoms during the past week (rated from 0 = none of the time to 4 = most of the time). The lowest score obtainable on the measure was 0, while the highest score obtainable was 76. Although no cut-off score was used, the higher the score on the scale, the greater the psychosocial distress being reported.
Time Frame: baseline, 3 week post-intervention and 6 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trauma-Focused Cognitive Behavioral Therapy | A Child Friendly Space
Number analyzed (Participants) | 26 | 24
units on a scale
  Pre-Intervention Scores | 45.08 (11.26) | 44.83 (9.25)
  Post-Intervention Scores | 19.04 (15.09) | 16.63 (9.36)
  6 month Follow-Up Intervention Scores | 12.77 (9.32) | 12.46 (8.54)

3. Secondary Outcome: Change in Externalizing Symptoms as Measured by the African Youth Psychosocial Assessment Instrument
Description: The African Youth Psychosocial Assessment Instrument is a self-report questionnaire that measures internalizing, externalizing, conduct and pro-social (daily life functioning) skills symptoms. The Congolese Swahili version of the AYPA contained 10 questions about symptoms of conduct disorder and assesses the frequency of occurrence of externalizing symptoms during the past week (rated from 0 = none of the time to 4 = most of the time). The lowest score obtainable on the measure was 0, while the highest score obtainable was 40. Although no cut-off score was used, the higher the score on the scale, the greater the psychosocial adjustment difficulties being reported.
Time Frame: baseline, 3-week post-intervention, 6-month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trauma-Focused Cognitive Behavioral Therapy | A Child Friendly Space
Number analyzed (Participants) | 26 | 24
units on a scale
  Pre-Intervention Scores | 13.88 (6.89) | 15.63 (6.54)
  Post-Intervention Scores | 5.35 (4.20) | 5.92 (4.41)
  6 month Follow-Up Intervention Scores | 4.35 (3.61) | 5.71 (5.39)

4. Secondary Outcome: Change in Pro-Social Behaviors as Measured by the African Youth Psychosocial Assessment Instrument
Description: The African Youth Psychosocial Assessment Instrument is a self-report questionnaire that measures internalizing, externalizing, conduct and pro-social (daily life functioning) skills symptoms. The Congolese Swahili version of the AYPA contained 8 questions about pro-social behavior and assesses the frequency of occurrence of positive behaviors (e.g. sharing with others, listening to others and elders etc.) during the past week (rated from 0 = none of the time to 4 = most of the time). The lowest score obtainable on the measure was 0, while the highest score obtainable was 32. Although no cut-off score was used, the higher the score on the scale, the more pro-social the individual's behavior is.
Time Frame: baseline, 3-week post-intervention, 6-month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trauma-Focused Cognitive Behavioral Therapy | A Child Friendly Space
Number analyzed (Participants) | 26 | 24
units on a scale
  Pre-Intervention Scores | 21.81 (5.84) | 22.96 (5.84)
  Post-Intervention Scores | 22.35 (3.86) | 23.33 (4.16)
  6 month Follow-Up Intervention Scores | 21.42 (4.24) | 18.75 (5.19)

ADVERSE EVENTS:
Arm/Group | Trauma-Focused Cognitive Behavioral Therapy | A Child Friendly Space
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No